CLINICAL TRIAL: NCT00420940
Title: The Effect of Daily Whole-Body Vibration on Tibial Trabecular Bone Mineral Density in Osteopenic Postmenopausal Women
Brief Title: The Influence of Vibration on Bone Mineral Density in Women Who Have Weak Bones After Menopause
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: PI - Dr. Angela M. Cheung, University Health Network/University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06-0332-AE; PSI 06-28 (Other Grant/Funding Number: The Physicians' Services Incorporated Foundation)
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2008-10

CONDITIONS: Bone Density; Osteopenia; Osteoporosis; Post-Menopause
Keywords: vibration; mechanical loading; bone mineral density; women's health; osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 90 Hz whole-body vibration (Experimental): 20-minute daily whole-body vibration at 90 Hz and 0.3g
  Interventions: Device: Juvent 1000 Dynamic Motion Therapy (DMT) Platform
- 30 Hz whole-body vibration (Experimental): 20-minute daily whole-body vibration at 90 Hz and 0.3g
  Interventions: Device: Juvent 1000 Dynamic Motion Therapy (DMT) Platform
- control (No Intervention): control group (receiving no vibration)

INTERVENTIONS:
Device: Juvent 1000 Dynamic Motion Therapy (DMT) Platform — Standing on a DMT whole-body vibration platform for 20 minutes per day at a frequency of 90 Hz and acceleration due to gravity of 0.3g
  Other Names: low magnitude whole-body vibration platform
  Arms: 90 Hz whole-body vibration
Device: Juvent 1000 Dynamic Motion Therapy (DMT) Platform — Standing on a DMT whole-body vibration platform for 20 minutes per day at a frequency of 90 Hz and acceleration due to gravity of 0.3g
  Other Names: low magnitude whole-body vibration platform
  Arms: 30 Hz whole-body vibration

SUMMARY:
This study will examine whether whole-body vibration slows down bone loss in healthy postmenopausal women with osteopenia. Whole-body vibration is a promising novel therapy that involves standing on a platform which produces extremely small and fast up-and-down movements. Some but not all research studies have found that whole-body vibration slowed down bone loss in postmenopausal women. One of the reasons why different studies found different results may be because they used various speeds of vibration. This study looks at how different speeds of whole-body vibration influence bone mineral density differently in postmenopausal women who have osteopenia. Two hundred postmenopausal women will take part in this 12-month study. Women will be randomly assigned into three groups (67 women per group) and these groups will be compared. Group 1 will receive very fast whole-body vibration, Group 2 will receive fast whole-body vibration, and Group 3 will not receive whole-body vibration. We will look at various bone mineral density and bone quality measurements, obtained with three different types of technologies, at the beginning of the study and at 12 months of follow-up. The hypothesis of this study is that the in comparison to Group 3 (no vibration), Groups 1 and 2 will experience reduced bone loss over 12 months, and that the greatest reduction in bone loss will be experienced by Group 1. The results of this study will help us determine whether whole-body vibration at different speeds produces variable effects on bone, hence explaining the inconsistency of the results obtained in previous studies.

DETAILED DESCRIPTION:
BACKGROUND:

Recent animal studies have shown that whole-body vibration increases bone mineral density. The effect of whole-body vibration on bone has been examined in only six small human studies with inconsistent results. Two of these studies have shown whole-body vibration reduces bone loss after menopause. Studies that used higher speed whole-body vibration may have produced greater reductions in bone loss.

OBJECTIVE AND HYPOTHESIS:

The objective of this study is to examine the effects of two whole-body vibration speeds trabecular BMD in the lower leg in osteopenic postmenopausal women. Two hundred postmenopausal women will take part in this 12-month study. Women will be randomly assigned into three groups (67 women per group) and these groups will be compared. Group 1 will receive very fast (90 Hz) whole-body vibration, Group 2 will receive fast (30 Hz) whole-body vibration, and Group 3 will not receive whole-body vibration. The hypothesis of this study is that the in comparison to Group 3 (no vibration), Groups 1 (very fast vibration, 90 Hz) and 2 (fast vibration, 30 Hz) will experience reduced bone loss over 12 months, and that the greatest reduction in bone loss will be experienced by Group 1.

METHODOLOGY:

Women with any clinical conditions that affect bone and those receiving drugs that affect bone will be excluded. The whole-body vibration therapy will involve standing barefoot and upright on a vibration platform daily for 20 minutes. Data will be collected at baseline, and at 12 months of follow-up. Our primary analysis will evaluate whether there are differences in changes in trabecular BMD in the lower leg (as measured by peripheral quantitative computed tomography; pQCT) between Groups 1, 2, and 3. Our secondary analyses will examine whether there are differences in changes in the following bone characteristics between Groups 1, 2, and 3:

1. trabecular bone quality in the lower leg (as measured by pQCT)
2. cortical bone BMD and quality in the lower leg (as measured by pQCT)
3. trabecular and cortical bone BMD and quality in the wrist (as measured by pQCT)
4. BMD at the hip and spine (as measured by dual x-ray absorptiometry, DXA)
5. BMD and quality at the heel (as measured by quantitative ultrasound).

SIGNIFICANCE:

Based on current scientific understanding of bone remodeling, vibration devices have the potential to play a significant part in maintaining bone health in postmenopausal women. The results of this study will help us determine whether low-magnitude, high-frequency WBV at different vibration rates produces variable effects on bone, hence explaining the inconsistency of the results obtained previously. This study will also lay the ground work for future large-scale randomized controlled trials that are needed to investigate the long-term effects of WBV on preventing postmenopausal bone loss. If effective, WBV can be another non-pharmaceutical strategy to decrease bone loss in postmenopausal women. This in turn will decrease the number of osteoporotic fractures and their associated morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* osteopenic
* postmenopausal

Exclusion Criteria:

* use of HRT in the past 12 months
* use of raloxifene or parathyroid hormone in the past 6 months
* use of bisphosphonates or fluoride in the past 3 months or ever taken for more than 3 months
* current use of calcitonin
* use of other medications that may indirectly affect bone metabolism
* presence of metabolic bone disease or diseases that indirectly affect bone metabolism
* occurrence of fragility fracture over 40 years of age
* presence of unhealed non-fragility fracture (i.e., occurring less then 6 months ago)
* having body mass ≤28 kg and ≥90 kg
* having knee or hip joint replacements and spine implants
* having poor balance (assessed by Timed-Up-and-Go)
* presence of other medical risks for the study
* inability to stand erect daily for 20 minutes
* planned vacation or other activities that would prevent one from using the platform for ≥1 month

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Trabecul volumetric bone mineral density (BMD) of the lower tibia (using peripheral quantitative computed tomography; pQCT)) | Baseline and 12 months

SECONDARY OUTCOMES:
Total BMD of the lower tibia (using pQCT) | Baseline and 12 months
Cortical BMD and cortical thickness of the lower tibia (using pQCT) | Baseline and 12 months
Trabecular thickness, separation, and number of the lower tibia (using pQCT) | Baseline and 12 months
Total BMD of the distal radius (using pQCT) | Baseline and 12 months
Cortical BMD and cortical thickness of the distal radius (using pQCT) | Baseline and 12 months
Trabecular BMD and thickness, separation, and number of the distal radius (using pQCT) | Baseline and 12 months
BMD at the total hip (using dual x-ray absorptiometry; DXA) | Baseline and 12 months
BMD at the femoral neck (using DXA) | Baseline and 12 months
BMD lumbar spine (using DXA) | Baseline and 12 months
BMD at the calcaneus (using quantitative ultrasound; QUS) | Baseline and 12 months
Speed of sound and broadband ultrasound attenuation at the calcaneus (QUS) | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Cheung, M.D., Ph.D., Principal Investigator — University Health Network, University of Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Slatkovska L, Alibhai SM, Beyene J, Hu H, Demaras A, Cheung AM. Effect of 12 months of whole-body vibration therapy on bone density and structure in postmenopausal women: a randomized trial. Ann Intern Med. 2011 Nov 15;155(10):668-79, W205. doi: 10.7326/0003-4819-155-10-201111150-00005. PMID 22084333